CLINICAL TRIAL: NCT05636566
Title: Comparison Between TIVA Using Propofol or Dexmedetomidine Versus Sevoflurane During Anaesthesia of Children Undergoing Bone-Marrow Aspiration
Brief Title: Comparing TIVA Using Propofol or Dexmedetomidine Versus Sevoflurane During Anaesthesia of Children Undergoing Bone-Marrow Aspiration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0305414
Record Dates: First submitted 2022-11-18; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-02

CONDITIONS: Invasive Cancer; Pediatric Cancer
Keywords: Dex-Profol; sevoflurane
MeSH Terms: conditions — Neoplasms | interventions — Sevoflurane; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Sixty patients were randomized and assigned into 3 groups (n=20) each, using sealed envelope technique:
  * Group (S): received sevoflurane- oxygen for induction and sevoflurane with fentanyl (Fentanyl, Janssen-Cilag, Germany) infusion for maintenance of anaesthesia.
  * Group (P): received propofol (Diprivan, Astra Zeneca, Wedel, Germany) for induction followed by propofol-fentanyl infusions for maintenance of anaesthesia.
  * Group (D): received dexmedetomedine (Precedex, Dexmedetomedine HCL inj.,Hospira, Inc.,Lacke Forest, USA) infusion for induction followed by dexmedetomedine-fentanyl infusions for maintenance of anaesthesia. All solutions were prepared by a team member not participating in data recording of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (S) (Active Comparator): sevoflurane inhalational anaesthesia for induction, then sevoflurane and fentanyl infusion for maintenance ,
  Interventions: Drug: Sevoflurane
- Group P (Active Comparator): propofol infusion for induction afterward propofol and fentanyl infusions for maintenance of anaesthesia
  Interventions: Drug: Propofol infusion for maintance
- Group D (Active Comparator): dexmedetomedine infusion for induction after that dexmedetomedine and fentanyl infusions for maintenance
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Sevoflurane — inhalational anaesthesia for maintenance
  Arms: Group (S)
Drug: Propofol infusion for maintance — propofol infusion after induction for maintenance of anaesthesia
  Arms: Group P
Drug: Dexmedetomidine — 0.5 mic /kg dexmedetomedine is injected after induction of anaesthesia
  Arms: Group D

SUMMARY:
No doubt that children facing surgical procedures are subjected to perioperative distressing, anxious and worrying periods. Several factors included; parental deprivation, anxiety, previously mismanaged experience and anticipating pain from the procedure itself weather diagnostic or curative. Anaesthetic goals should focus at alleviating these unfavorable events that may exacerbate the inevitable associated neurohormal stress response with its injurious effects on the course of the procedure. Moreover, it likely to extend beyond the surgical procedure predisposing these vulnerable group of patients to psychological trauma and chronic behavioral changes.

Bone marrow aspiration (BMA) is a frequent procedure that necessitate a meticulous anaesthetic plane that entails rapid non-traumatic induction together with adequate pain free maintenance and instant smooth recovery after a short time practice. Total intravenous anaesthesia (TIVA) had emerged as alternative anaesthetic technique to inhalational anaesthesia for conscious sedation in BMA cited by many authors.

Propofol a popular anaesthetic/ sedative with a rapid onset, short duration and smooth recovery of consciousness and psychomotor functions with no cumulation. However it is poorly analgesic, depresses respiration and there is a possibility of loss of muscle tone leading to airway obstruction .

Dexmedetomidine is a greatly active α2 adrenergic agonist with a valuable anaesthetic- analgesic saving effects. It augments sedation, hypnosis and preservation of muscle tone with negligible respiratory depression and hemodynamic derangements.

The purpose of the current study is to compare between effects of TIVA using propofol or dexmedetomedine versus sevoflurane for maintenance of anaesthesia in children undergoing bone marrow aspiration.

DETAILED DESCRIPTION:
Background: although bone marrow aspiration in children is a familiar short duration procedure, nearly 65% of patients develop sever anxiety that may extend more beyond, up to chronic postoperative behavioral changes. Consequently, the objectives of any related anaesthetic technique is to afford smooth non-traumatic induction with safe maintenance and rapid recovery. The rational of the present study is to compare between TIVA using propofol or dexmedetomedine and sevoflurane for maintenance of anaesthesia in children scheduled for bone marrow aspiration.

Patients and methods: 60 child aged 3-12 years with ASA physical status I and II planned for elective bone marrow biopsy and aspiration were enrolled randomly into 3 groups 20 child each; group(S): received sevoflurane- oxygen for induction and sevoflurane with fentanyl infusion for maintenance of anaesthesia. Group (P): received propofol for induction followed by propofol-fentanyl infusions for maintenance of anaesthesia. Group (D): received dexmedetomedine infusion for induction followed by dexmedetomedine-fentanyl infusions for maintenance of anaesthesia. The primary endpoint was postoperative sedation score on arrival to the post anaesthetic care unit (PACU) after surgery. Secondary outcomes included procedure duration, hemodynamic variables, parents and surgeons satisfaction and incidences of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 3-12 years.
* both sexes
* ASA physical status I and II

Exclusion Criteria:

* Patients with identified allergy to the study medications
* with recognized lipid or carbohydrate deranged metabolism
* cardiac dysrhythmias
* congenital heart diseases
* cardiomyopathy
* significant organ dysfunction.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
sedation score | immediately postoperative
  indicator for post operative alertness, . Sedation level: Agitated = 4, Awake= 3, Drowsy= 2, Asleep= 1. A sedation score of 3 & above was considered as unsatisfactory while 1 & 2 is considered to be satisfactory.

SECONDARY OUTCOMES:
time for spontenous eye opening | immediately postoperative
  assessement of the immediate time of recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicin, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No